CLINICAL TRIAL: NCT03822377
Title: Ticagrelor Administered as Standard Tablet or orodispersiblE foRmulation
Acronym: TASTER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Azienda Ospedaliero Universitaria di Sassari (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Prof. Guido Parodi, Professor, Azienda Ospedaliero Universitaria di Sassari
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ESR-17-13174; 2018-001790-25 (EudraCT Number)
Record Dates: First submitted 2019-01-23; First posted 2019-01-30 (Actual); Results first posted 2021-09-08 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: ST Elevation Myocardial Infarction; NSTEMI - Non-ST Segment Elevation MI
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: Comparison of platelet inhibition at different timepoints between 65 patients in the treatment arm (receiving orodispersible formulation of ticagrelor loading dose) versus 65 patients in the control arm (receiving standard coated formulation of ticagrelor loading dose). Randomization will be further stratified according to morphine use.
Who Masked: Investigator
Masking Description: Site investigators performing platelet function tests will be blinded regarding patient randomization arm and the blood samples will be fully anonymized.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ticagrelor orodispersible tablets (Experimental): STEMI or very high-risk NSTEMI patients undergoing primary PCI and receiving Ticagrelor 180 mg loading dose as orodispersible tablets.
  Intervention: administration of Ticagrelor 180 mg loading dose as orodispersible tablets.
  Interventions: Drug: Ticagrelor orodispersible tablets
- Ticagrelor standard tablets (Active Comparator): STEMI or very high-risk NSTEMI patients undergoing primary PCI and receiving Ticagrelor 180 mg loading dose as standard coated tablets.
  Intervention: administration of Ticagrelor 180 mg loading dose as standard coated pills.
  Interventions: Drug: Ticagrelor standard tablets

INTERVENTIONS:
Drug: Ticagrelor orodispersible tablets — Ticagrelor loading dose (180 mg) given as two orodispersible tablets (each of 90 mg), to be dispersed in saliva.
  Arms: Ticagrelor orodispersible tablets
Drug: Ticagrelor standard tablets — Ticagrelor loading dose (180 mg) given as two standard coated tablets (each of 90 mg) to be swallowed with water.
  Arms: Ticagrelor standard tablets

SUMMARY:
Randomized clinical study evaluating superiority in platelet inhibition after administration of Ticagrelor 180 mg loading dose as an orodispersible formulation versus traditional coated tablets in patients admitted for ST elevation myocardial infarction or very high-risk non-ST elevation myocardial infarction.

DETAILED DESCRIPTION:
Primary percutaneous coronary intervention (PPCI) is the preferred reperfusion strategy for patients with acute ST-segment elevation myocardial infarction (STEMI). Additional antithrombotic therapy prior or during intervention plays an important role in the short- and long-term outcomes after PPCI. Oral antiplatelet therapy including a platelet P2Y12 receptor inhibitors is a cornerstone of antithrombotic treatment in patients with acute coronary syndromes. Prasugrel and Ticagrelor have been shown to be superior to Clopidogrel in patients with STEMI in reduction of ischemic complication without any increase in the bleeding risk and with a significant reduction in the stent thrombosis rate. Nevertheless, in STEMI patients, pharmacodynamic studies showed prasugrel and ticagrelor oral loading dose (LD) provided a suboptimal platelet inhibition in the first hours after LD, and at least 4 hours are required to achieve and effective platelet aggregation inhibition in the majority of patients, in part due to slowed gut motility caused by morphine use. Orodispersible tablet (ODT) is a different tablet formulation that disperses upon contact with the moist mucosal surfaces of the oral cavity and quickly release its components before swallowing; thus local drug dissolution and absorption as well as onset of clinical effect can be obtained conveniently easily and quickly by bypassing gastrointestinal tract. Recently, Ticagrelor 90 mg ODT has become available and bioequivalence studies on healthy volunteers documented its effectiveness with consequent approval by European Medicine Agency of this formulation which is currently available on the market. Thus, the aim of the present study is to evaluate the superiority in platelet inhibition with 180 mg Ticagrelor loading dose (LD) administered as ODTs as compared with standard formulation, among patients with STEMI or very high-risk NSTEMI undergoing immediate PCI. Primary objective consists in evaluating platelet reactivity 1 hour after Ticagrelor loading dose by VerifyNow test.

ELIGIBILITY:
Inclusion Criteria:

1. Patients presenting within 12 hours from the onset of symptoms with STEMI or very high-risk NSTEMI referred for immediate (< 2 hours) angiography. Very high-risk NSTEMI patients include patients with haemodynamic instability or cardiogenic shock, heart failure, life-threatening arrhythmias or resuscitated cardiac arrest, intermittent ST-segment elevation, or ongoing chest pain.
2. Informed, written consent
3. Male or female patients, aged ≥ 18 years old

Exclusion Criteria:

1. Age < 18 years
2. Active bleeding; bleeding diathesis; coagulopathy
3. History of gastrointestinal or genitourinary bleeding <2 months
4. Major surgery in the last 6 weeks
5. History of intracranial bleeding or structural abnormalities
6. Suspected aortic dissection
7. Administration in the week before the index event of clopidogrel, ticlopidine, prasugrel, ticagrelor, thrombolytics, bivalirudin, low-molecular weight heparin or fondaparinux.
8. Concomitant oral or IV therapy with strong CYP3A inhibitors or strong CYP3A inducers, CYP3A with narrow therapeutic window
9. Known relevant hematological deviations: Hb <10 g/dl, Thromb. <100x10^9/l
10. Use of warfarin or new oral anticoagulant derivatives within the last 7 days
11. Known severe liver disease, severe renal failure
12. Allergy or hypersensitivity to ticagrelor or any of the excipients.
13. Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2019-06-27 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guido Parodi, Professor, Principal Investigator — Cardiologia Clinica e Interventistica - AOU Sassari
Locations (1):
- Cardiologia Clinica e Interventistica - AOU Sassari, Sassari, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Parodi G, Talanas G, Mura E, Canonico ME, Siciliano R, Guarino S, Marini A, Dossi F, Franca P, Raccis M, Saba PS, Sanna GD. Orodispersible Ticagrelor in Acute Coronary Syndromes: The TASTER Study. J Am Coll Cardiol. 2021 Jul 20;78(3):292-294. doi: 10.1016/j.jacc.2021.05.015. No abstract available. PMID 34266583

RESULTS

PARTICIPANT FLOW:
Groups:
- Ticagrelor Orodispersible Tablets: STEMI or very high-risk NSTEMI patients undergoing primary PCI and receiving Ticagrelor 180 mg loading dose as orodispersible tablets.
  Intervention: administration of Ticagrelor 180 mg loading dose as orodispersible tablets.
  Ticagrelor orodispersible tablets: Ticagrelor loading dose (180 mg) given as two orodispersible tablets (each of 90 mg), to be dispersed in saliva.
- Ticagrelor Standard Tablets: STEMI or very high-risk NSTEMI patients undergoing primary PCI and receiving Ticagrelor 180 mg loading dose as standard coated tablets.
  Intervention: administration of Ticagrelor 180 mg loading dose as standard coated pills.
  Ticagrelor pills: Ticagrelor loading dose (180 mg) given as two standard coated tablets (each of 90 mg) to be swallowed with water.
Period: Overall Study
Arm/Group | Ticagrelor Orodispersible Tablets | Ticagrelor Standard Tablets
Started | 65 | 65
Completed | 65 | 65
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ticagrelor Orodispersible Tablets | Ticagrelor Standard Tablets | Total
Number analyzed (Participants) | 65 | 65 | 130
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.0 (10.0) | 63.0 (10.0) | 63.5 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 17 | 25
  Male | 57 | 48 | 105
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 65 | 65 | 130
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of Platelet Inhibition
Description: Platelet reactivity will be measured by VerifyNow test 1 hour after Ticagrelor loading dose (LD) administered as orodispersible tablets as compared with standard formulation in 130 patients with STEMI or very high-risk NSTEMI undergoing immediate PCI.
  The VerifyNow PRU Test is designed to measure P2Y12 receptor blockade. Results of the PRU Tests are reported as P2Y12 Reaction Units (PRU). PRU measures the extent of platelet aggregation in the presence of a P2Y12 inhibitor. Lower PRU levels are associated with expected antiplatelet effect.
Time Frame: 1 hour
Measure: Median (Inter-Quartile Range); unit: P2Y12 Reaction Units (PRU)
Arm/Group | Ticagrelor Orodispersible Tablets | Ticagrelor Standard Tablets
Number analyzed (Participants) | 65 | 65
P2Y12 Reaction Units (PRU) | 94 [35 to 193] | 141 [8 to 197]

2. Secondary Outcome: Percent of Patients With Insufficient Antiaggregation
Description: The percent of patients with a high residual platelet reactivity (PRU > 208 by VerifyNow test), thus not adequately antiaggregated, 1 hour after Ticagrelor LD.
Time Frame: 1 hour
Measure: Count of Participants; unit: Participants
Groups:
- Experimental Arm: STEMI or very high-risk NSTEMI patients undergoing primary PCI and receiving Ticagrelor 180 mg loading dose as orodispersible tablets.
  Intervention: administration of Ticagrelor 180 mg loading dose as orodispersible tablets.
  Ticagrelor orodispersible tablets: Ticagrelor loading dose (180 mg) given as two orodispersible tablets (each of 90 mg), to be dispersed in saliva.
- Control Arm: STEMI or very high-risk NSTEMI patients undergoing primary PCI and receiving Ticagrelor 180 mg loading dose as standard coated tablets.
  Intervention: administration of Ticagrelor 180 mg loading dose as standard coated pills.
  Ticagrelor pills: Ticagrelor loading dose (180 mg) given as two standard coated tablets (each of 90 mg) to be swallowed with water.
Arm/Group | Experimental Arm | Control Arm
Number analyzed (Participants) | 65 | 65
Participants | 51 | 53

3. Secondary Outcome: Number of Participants With Residual Platelet Reactivity at Various Timepoints
Description: Residual platelet reactivity (PRU) at 2, 4 and 6 hours measured by VerifyNow test to assess antiplatelet effect of P2Y12 inhibitors
Time Frame: 2, 4 and 6 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Ticagrelor Orodispersible Tablets | Ticagrelor Standard Tablets
Number analyzed (Participants) | 65 | 65
Participants | 42 | 9

4. Secondary Outcome: Number of Participants With Clinically Relevant Bleeding Events
Description: Actionable bleeding events across the two different regimens of Ticagrelor administration, requiring diagnostic studies, hospitalization, or treatment by a health care professional (BARC type 2 or higher)
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Ticagrelor Orodispersible Tablets | Ticagrelor Standard Tablets
Number analyzed (Participants) | 65 | 65
Participants | 0 | 4

5. Other Pre Specified Outcome: Number of Participants With Morphine-ticagrelor Interaction
Description: Potential morphine-ticagrelor interaction will be assessed by stratified randomization according to morphine use
Time Frame: 6 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Ticagrelor Orodispersible Tablets | Ticagrelor Standard Tablets
Number analyzed (Participants) | 65 | 65
Participants | 6 | 4

6. Other Pre Specified Outcome: Incidence of Adverse Events Occurring During Hospital Stay
Description: Combined ticagrelor administration-related adverse events defined as in-hospital ≥2 BARC bleedings, dyspnea, ventricular pauses, allergic reactions, or vomit
Time Frame: Until discharge from the hospital (usually up to 7 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Arm | Control Arm
Number analyzed (Participants) | 65 | 65
Participants | 14 | 15

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Ticagrelor Orodispersible Tablets | Ticagrelor Standard Tablets
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/65
Serious Adverse Events (participants affected / at risk) | 1/65 | 0/65
Other Adverse Events (participants affected / at risk) | 14/65 | 15/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ticagrelor Orodispersible Tablets (N=65) | Ticagrelor Standard Tablets (N=65)
Reinfarction (Cardiac disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ticagrelor Orodispersible Tablets (N=65) | Ticagrelor Standard Tablets (N=65)
Combined ticagrelor administration-related adverse events defined as in-hospital ≥2 BARC bleedings, (Cardiac disorders) | 14 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-07): https://cdn.clinicaltrials.gov/large-docs/77/NCT03822377/Prot_SAP_000.pdf